CLINICAL TRIAL: NCT03443141
Title: Effecto of Total Occlusive Vitamin E-containing Dressing on Incisional Surgical Site Infection in Elective Laparoscopic Colorectal Surgery
Brief Title: Effect of Vitamin E-containing Dressing on Surgical Site Infection in Colorectal Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Professor of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HRJC2018-20
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Vitamin E; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin E dressing (Experimental): Patients will receive a Vitamin E-containing dressing over the wound
  Interventions: Drug: Vitamin E
- Standard dressing (Sham Comparator): Patients will receive a standard dressing over the wound
  Interventions: Drug: Standard dressing

INTERVENTIONS:
Drug: Vitamin E — The applied dressing will be embebbed in Vitamin E
  Other Names: Exerimental group
  Arms: Vitamin E dressing
Drug: Standard dressing — The applied dressing is a normal one without adding any product to it.
  Other Names: Control group
  Arms: Standard dressing

SUMMARY:
A prospective, randomized study will be performed. Patients are randomized using a 1:1 allocation into 2 groups: patients receiving a vitamin E-containing dressing (group 1) and a conventional dressing (group 2). The primary outcomes variable will be occurrence of incisional SSI. Follow-up will be 30 days postoperatively.

DETAILED DESCRIPTION:
A prospective, randomized study will be performed. Patients are randomized using a random number table into 1:1 allocation into 2 groups: patients receiving a vitamin E-containing dressing (group 1) and a conventional dressing (group 2). In group 1 the wound will be covered with a Vitamin E embebbed gauze and plastic adhesive tape. In Group 2, , the wound will be covered with standard gauze and plastic adhesive tape.

The primary outcomes variable will be occurrence of incisional SSI, defined by CDC criteria. Follow-up will be 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of colorectal neoplasms
* plan to undergo an elective operation with curative aims
* laparoscopic surgery

Exclusion Criteria:

* Anastomotic leak
* Lost to 30-days follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Incisional surgical site infection | 30 days postoperatively
  Patients present a wound with the CDC criteria for SSI

CONTACTS AND LOCATIONS:
Overall Officials: Damian Garcia-Olmo, MD, PhD, Study Director — HOSPITAL REY JUAN CARLOS
Locations (1):
- Hospital general Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided